CLINICAL TRIAL: NCT05709626
Title: PRasugrEl Monotherapy Following prImary percUtaneous Coronary Intervention for ST-elevation Myocardial Infarction
Acronym: PREMIUM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kindai University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y0140
Record Dates: First submitted 2023-01-19; First posted 2023-02-02 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: Acute Coronary Syndrome; Dual AntiPlatelet Therapy; Drug Eluting Stent; Percutaneous Coronary Intervention; ST-elevation myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Acute Coronary Syndrome | interventions — N-acetyl-S-(alpha-methyl-4-(2-methylpropyl)benzeneacetyl)cysteine 4-(nitrooxy)butyl ester; 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No aspirin (Prasugrel monotherapy) (Active Comparator): To start prasugrel monotherapy before primary percutaneous coronary intervention (PCI).
  Interventions: Drug: No aspirin (Prasugurel monotherapy)
- 12-month DAPT (Active Comparator): To start dual antiplatelet therapy with prasugrel and aspirin for 12 months before primary percutaneous coronary intervention (PCI).
  Interventions: Drug: 12-month DAPT

INTERVENTIONS:
Drug: No aspirin (Prasugurel monotherapy) — 12-month prasugrel monotherapy
  Other Names: Experimental arm
  Arms: No aspirin (Prasugrel monotherapy)
Drug: 12-month DAPT — 12-month dual antiplatelet therapy with prasugrel and aspirin
  Other Names: Reference arm
  Arms: 12-month DAPT

SUMMARY:
The aim of this study is to evaluate the safety of prasugrel monotherapy without aspirin versus 12-month dual antiplatelet therapy (DAPT) in patients with STEMI using platinum-chrome everolimus-eluting stent (PtCr-EES: SYNERGYTM).

DETAILED DESCRIPTION:
In the STOPDAPT-2 ACS trial (NCT03462498), ischemic events (especially myocardial infarction) was significantly increased with 1-month DAPT followed by clopidogrel monotherapy, as compared to 12-month DAPT in patients with acute coronary syndrome (ACS). This was potentially attributable to clopidogrel, instead of prasugrel, which is more potent and has less individual difference in efficacy. On the other hand, previous studies including the STOPDAPT-2 ACS that evaluated the safety and efficacy of monotherapy with a P2Y12 inhibitor without aspirin consistently and significantly reduced the risk of bleeding, compared with standard DAPT. Consequently, there has been growing necessity to establish the safety with P2Y12 inhibitor monotherapy in terms of major adverse cardiovascular events. Therefore, we have planned to evaluate the non-inferiority of P2Y12 inhibitor monotherapy with prasugrel versus standard 12-month DAPT with prasugrel and aspirin in terms of the incidence of major cardiovascular events at 12 months after primary PCI in patients with STEMI using Platinum-Chromium Everolimus Eluting Stent (PtCr-EES; SYNERGYTM).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary PCI with everolimus-eluting stent (PtCr-EES, SYNERGYTM)
* STEMI patients
* Patients who can continue dual antiplatelet therapy with aspirin and a P2Y12 inhibitor for 12 months

Exclusion Criteria:

* Patients taking anticoagulants
* Patients under 18 years old
* Patients with less than 1 year prognosis
* Patients participating in other intervention studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2258 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2025-01-04 (Estimated); Study Completion 2028-01-04 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  Composite of all-cause death, myocardial infarction, or stroke

SECONDARY OUTCOMES:
Major secondary bleeding endpoint: Type 3 or 5 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 3 or 5 bleeding defined by BARC criteria
All-cause death | 12 months
  Death from any cause
Cardiovascular death | 12 months
  Death from cardiovascular cause
Non-cardiovascular death | 12 months
  Death from non-cardiovascular cause
Myocardial infarction (Periprocedual/ Spontaneous) | 12 months
  Defined by the Academic Research Consortium (ARC)-2
Stroke (Ischemic/ Haemorrhagic) | 12 months
  Including both ischemic and haemorrhagic stroke
Ischemic stroke | 12 months
  Ischemic stroke with symptom lasting over 24 hours
Hemorrhagic stroke | 12 months
  Intracerebral hemorrhage or subarachnoidal hemorrhage not associated with trauma
Stent thrombosis | 12 months
  Stent thrombosis defined by Academic Research Consortium (ARC)-2 definition
Target lesion failure | 12 months
  Cardiovascular death, target vessel myocardial infarction, clinically indicated target lesion revascularization
Target vessel failure | 12 months
  Cardiovascular death, target vessel myocardial infarction, clinically indicated target vessel revascularization
Patient-Oriented Composite Endpoint | 12 months
  All-cause death, stroke, myocardial infarction, and all revascularization, defined by the Academic Research Consortium (ARC)-2
Any target lesion revascularization | 12 months
  Revascularization to the target lesions (including 5mm of both ends of the stent[s]) regardless of PCI or CABG
Clinically-driven target lesion revascularization | 12 months
  Target lesion revascularization with the anginal symptoms or the positive test for ischemia
Non-target lesion revascularization | 12 months
  Revascularization to non-target lesions regardless PCI or CABG
Coronary artery bypass grafting | 12 months
  Any coronary artery bypass grafting
Any target vessel revascularization | 12 months
  Revascularization to the target vessel
Any coronary revascularization | 12 months
  Revascularization regardless of PCI or CABG
Type 2 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 2 bleeding defined by BARC criteria
Type 3 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 3 bleeding defined by BARC criteria
Type 4 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 4 bleeding defined by BARC criteria
Type 5 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 5 bleeding defined by BARC criteria
Type 2, 3, or 5 bleeding in Bleeding Academic Research Consortium (BARC) criteria | 12 months
  Type 2, 3, or 5 bleeding defined by BARC criteria
Major bleeding in Thrombolysis in Myocardial Infarction (TIMI) criteria | 12 months
  Major bleeding defined by TIMI criteria
Minor bleeding in Thrombolysis in Myocardial Infarction (TIMI) criteria | 12 months
  Minor bleeding defined by TIMI criteria
Major or minor bleeding in Thrombolysis in Myocardial Infarction (TIMI) criteria | 12 months
  Major or minor defined by TIMI criteria
Severe bleeding in Global utilization of streptokinase and tPA for occluded arteries (GUSTO) criteria | 12 months
  Severe bleeding defined by GUSTO criteria
Moderate bleeding in Global utilization of streptokinase and tPA for occluded arteries (GUSTO) criteria | 12 months
  Moderate bleeding defined by GUSTO criteria
Moderate or severe bleeding in Global utilization of streptokinase and tPA for occluded arteries (GUSTO) criteria | 12 months
  Moderate or severe bleeding defined by GUSTO criteria
Intracranial bleeding | 12 months
  Intracranial bleeding regardless of spontaneous or trauma
Gastrointestinal bleeding | 12 months
  Bleeding from gastrointestinal tract regardless of severity
Gastrointestinal complaints | 12 months
  Requirement of upper gastric fiberscopy to examine the gastrointestinal complaints

CONTACTS AND LOCATIONS:
Overall Officials: Gaku Nakazawa, MD, PhD, Principal Investigator — Kindai University Faculty of Medicine
Locations (1):
- Kindai University Faculty of Medicine, Sayama, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takahashi K, Kozuma K, Morino Y, Kashiwabara K, Otake H, Suwa S, Nanasato M, Muramatsu T, Anzai H, Shirakabe A, Yamamoto M, Asaumi Y, Sakuma M, Okayama H, Ikari Y, Nakazawa G. Prasugrel monotherapy versus 12-month dual antiplatelet therapy in STEMI patients undergoing intravascular imaging-guided PCI: Study design and rationale of the randomized PREMIUM trial. Cardiovasc Revasc Med. 2025 Dec 11:S1553-8389(25)00611-6. doi: 10.1016/j.carrev.2025.12.007. Online ahead of print. PMID 41436299